CLINICAL TRIAL: NCT00462124
Title: One-arm, Multi-center, Prospective Study to Assess the Safety and Efficacy of BioProtect Biodegradable Implantable Balloon in Prostate Cancer Subjects Undergoing Radiotherapy
Brief Title: Evaluation of the Safety and Efficacy of the BioProtect Balloon in Prostate Cancer Subjects Undergoing Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioProtect (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BP-01
Record Dates: First submitted 2007-04-16; First posted 2007-04-18 (Estimated); Results first posted 2019-08-08 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2018-02

CONDITIONS: Prostate Cancer
Keywords: Prostate; cancer; radiation; biodegradable implantable balloon; intrarectal balloon
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Balloon (Other): Implantation of a biodegradable balloon spacer (absorbable perirectal spacer)
  Interventions: Device: Absorbable perirectal spacer

INTERVENTIONS:
Device: Absorbable perirectal spacer — biodegradable balloon implant to increase the distance between prostate and anterior rectal wall

SUMMARY:
Primary Goal The study's primary goal is to assess the safety of the BioProtect biodegradable balloon implant and implantation procedure, in prostate cancer subjects undergoing routine XRT treatment. Safety of the BioProtect device will be assessed by reporting adverse events.

Secondary Goal The study's secondary goal is to evaluate the effectiveness of the BioProtect biodegradable balloon implant in prostate cancer subjects undergoing routine XRT treatment. Effectiveness will be assessed in terms of increased distance between anterior rectal wall and prostate and noticeable reduction of isodose to the rectum.

DETAILED DESCRIPTION:
Primary Endpoint Parameters

The safety endpoint is incidence of complications related to BioProtect balloon implant and implantation procedure:

1. Serious Adverse Events related to the BioProtect balloon and/or implantation procedure. Serious adverse event are defined as adverse requiring operation and/or associated with prolongation of hospital stay. Serious Adverse Events will be documented in Serious Adverse Event Form.
2. Adverse Events related to the BioProtect balloon and/or implantation procedure. Adverse Events will be documented in Adverse Event Form.
3. Subjective discomfort related to the balloon and implantation procedure will be assessed by pain analogue scale.

Secondary Endpoint Parameters

To assess the efficacy of BioProtect biodegradable balloon implant. Efficacy will be measured in terms of:

1. Increased distance between anterior rectal wall and prostate post implantation as showed by CT until last radiation treatment.
2. Noticeable reduction of isodose level to the rectum post implantation as compared to pre-implantation isodose to the rectum by XRT treatment planning software.

Other Measured Observations

1. Balloon non-displacement during treatment phase as shown by CT.
2. Balloon remaining inflated during treatment phase as shown by CT.
3. Operator satisfaction from BioProtect balloon implantation procedure.

ELIGIBILITY:
Inclusion Criteria:

* Male aged ≤80.
* Men with child producing potential (that are not sterile) must accept using adequate contraceptive throughout the radiotherapy phase and for at least 3 months after completion of the radiotherapy phase when ever they have heterosexual intercourse.
* Diagnosed prostate cancer not spread outside the capsule (T1 and T2).
* Subject is scheduled for localized prostate XRT treatments.
* Zubrod performance status 0-1; or Karnofsy >80.
* Pre-randomization serum PSA lower than 25 (obtained prior to any LHRH or antiandrogen therapy); or Kattan nomogram less than 15 %.
* Subject able to comprehend and give informed consent for participation in this study.
* Probability of lymph node involvement based on Kattan nomogram less than 15 %.
* Normal blood CBC and biochemistry up to two weeks before screening as follow:

  * Normal CBC
  * Absolute neutrophil count (ANC) ≥ 1,800 cells/mm3
  * Platelets ≥ 100,000 cells/mm3
  * Hemoglobin ≥ 10.0 g/dl
  * Adequate renal function, with serum creatinine ≤ 2.0 mg/dl
  * Adequate liver function, with serum bilirubin < 2.0 mg/dl
  * Adequate liver function with SGOT/SGPT < 2.5 x the upper normal limit
  * Normal values of the PT, PTT and INR tests.
* Signed Informed Consent Form.

Exclusion Criteria:

* Prior radical prostatectomy, cryosurgery or radiotherapy for prostate cancer, or other local therapy for prostate cancer.
* Prior radiotherapy to the pelvis, including brachytherapy at the same body organ.
* Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months prior to screening.
* Transmural myocardial infarction within the last 6 months prior to screening.
* Acute infection requiring intravenous antibiotics at the time of screening.
* Bleeding disorders.
* Uncontrolled diabetes mellitus
* HIV positive or any other immunosuppressive disorder.
* Renal failure (Serum creatinine >2.0 mg/dl).
* Inflammatory diseases of the perineal skin.
* Urinary tract infection or acute or chronic prostatitis.
* Active inflammatory bowel disease.
* Rectal carcinoma.
* Subjects after anterior resection of rectum or after rectal amputation.
* Known cognitive disorder.
* Concurrent participation in any other clinical study.
* Physician objection.

Max Age: 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-06; Primary Completion 2009-03 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yossi Muncher, Dr., Study Director — BioProtect
Locations (1):
- Ichilov Medical Center, Tel Aviv, Israel

RESULTS

PARTICIPANT FLOW:
Groups:
- Balloon Implant: Absorbable perirectal spacer implantation
Period: Overall Study
Arm/Group | Balloon Implant
Started | 7
Completed | 6 (One implant was misplaced and was disacitivated by puncture.)
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Balloon Implant: Implantation of a biodegradable balloon spacer (absorbable perirectal spacer) to increase the distance between prostate and anterior rectal wali.
Arm/Group | Balloon Implant
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 7
Region of Enrollment [Number; unit: participants]
  Israel | 7

OUTCOME MEASURES:

1. Primary Outcome: Safety of Balloon Implant
Description: Assessed by collecting number of subjects experiencing a serious device related adverse event.
Time Frame: 6 months
Population: ITT
Measure: Number; unit: Participants
Arm/Group | Balloon Implant
Number analyzed (Participants) | 7
Participants | 0

2. Secondary Outcome: Efficacy Will be Measured in Terms of: Number of Participants With a Reduction in Radiation to the Rectum
Description: The space between the prostate and the rectum will be determined by Ct in subjects with prostate cancer who underwent radiotherapy and who received the balloon. The degree of increase in this space is directly related to a reduction of isodose level delivered to the rectum, and therefore a reduction in post radiation therapy rectal adverse event sequela.
Time Frame: 6 months
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Balloon Implant
Number analyzed (Participants) | 7
Participants | 7

ADVERSE EVENTS:
Time Frame: 13 months
Description: Rectal perforation was considered serious, even if no symptoms develop nor sequela arise.
Groups:
- Group 1: Absorbable perirectal spacer implantation
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 1/7
Other Adverse Events (participants affected / at risk) | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=7)
Tear in rectal mucosa (Gastrointestinal disorders) | 1 (1) — Due to anatomical adhesions, rectal mucosa was flattened during inflation and caused rectal mucosal tear which did not penetrate to inner wall. Previous treatment in the area was excluded in future studies. Physician did not consider event serious.
Urinary retention (Renal and urinary disorders) | 1 (1) — Due to previous surgery, the urethra was pressued by the balloon and caused urinary retention and the subject was hospitalized.

LIMITATIONS AND CAVEATS:
This was an initial human experience feasibility study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No